CLINICAL TRIAL: NCT01187823
Title: Comparison of Adaptive Servo Ventilation(Bipap® Auto SV Advanced) and Oxgen Therapy in Chronic Heart Failure Patients Complicated With Central Sleep Apnea
Brief Title: The Effect of Adaptive Servo Ventilation and Oxygen Therapy in Central Sleep Apnea Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyoto University, Graduate School of Medicine (Other)
Collaborators: Philips Respironics (Industry); Philips Healthcare (Industry)
Responsible Party: Principal Investigator, Kimihiko Murase, medical doctor, Kyoto University, Graduate School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-447
Record Dates: First submitted 2010-08-23; First posted 2010-08-24 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Heart Failure; Sleep Apnea
Keywords: Chronic heart failure; Central sleep apnea; Obstructive sleep apnea; Adaptive servo ventilation
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Central; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nocturnal oxygen therapy (Active Comparator)
  Interventions: Device: Nocturnal oxygen
- Adaptive servo ventilation (Active Comparator): Bipap® auto SV Advanced
  Interventions: Device: Adaptive servo ventilation

INTERVENTIONS:
Device: Adaptive servo ventilation — Nocturnal use of Adaptive servo ventilation
  Other Names: Bipap® auto SV Advanced (Philips Respironics)
  Arms: Adaptive servo ventilation
Device: Nocturnal oxygen — Nocturnal use of oxygen
  Arms: Nocturnal oxygen therapy

SUMMARY:
The aim of this study is to compare the effects of Adaptive Servo Ventilation (Bipap® auto SV Advanced) and oxygen therapy in chronic heart failure patients complicated with central sleep apnea.

DETAILED DESCRIPTION:
Central sleep apnea(CSA) is associated with chronic heart failure(CHF). At present, both of nocturnal oxygen therapy and adaptive servo ventilation(ASV) are recognized as effective modalities. However,in fact, majority of CHF patients are complicated not only with CSA but with obstructive sleep apnea(OSA). Recently, Philips developed Bipap® auto SV Advanced for such patients. It has auto-CPAP function as the modality of OSAS, in addition to ASV function. The present study is prospective randomised study to compare the effects of nocturnal oxygen therapy and Bipap® auto SV Advanced.

ELIGIBILITY:
Inclusion Criteria:

* Left ventricular ejection fraction<50% confirmed by echocardiography
* Apnea hypopnea index(AHI)>=20 confirmed by overnight polysomnography
* More than 15% of AHI is due to CSA

Exclusion Criteria:

* Changes of cardioactive drug prescriptions within 6 weeks
* Admission due to cardiovascular events within 6 weeks
* Ever used CPAP or ASV for sleep apnea
* Ever used nocturnal oxgen therapy
* Subjects with acute exacerbation of chronic heart failure
* Operation for upper airway within 90 days
* Renal dialysis
* History of stroke with neurological deficit

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction confirmed by echocardiography | three months

SECONDARY OUTCOMES:
Sleep quality confirmed by polysomnography | three months
Endothelial function | three months
Sleepiness | three months
Blood pressure | three months
Serum biomarkers | three months
  Inflammation, oxidative stress
health-related quality of life | three months
Urinary biomarkers | three months
  inflammation, oxidative stress
Heart rate | three months

CONTACTS AND LOCATIONS:
Overall Officials: Kazuo Chin, MD, PhD, Principal Investigator — Kyoto University, Graduate School of Medicine; Takeshi Kimura, MD,PhD, Principal Investigator — Kyoto University, Graduate School of Medicine; MIchiaki Mishima, MD,PhD, Study Chair — Kyoto University, Graduate School of Medicine; Kimihiko Murase, MD, Principal Investigator — Kyoto University, Graduate School of Medicine
Locations (1):
- Kyoto University Hospital, Kyoto, Kyoto, Japan

REFERENCES:
- [Derived] Murase K, Ono K, Yoneda T, Iguchi M, Yokomatsu T, Mizoguchi T, Izumi T, Akao M, Miki S, Nohara R, Ueshima K, Mishima M, Kimura T, White DP, Chin K. Adaptive servoventilation versus oxygen therapy for sleep disordered breathing in patients with heart failure: a randomised trial. Open Heart. 2016 Mar 31;3(1):e000366. doi: 10.1136/openhrt-2015-000366. eCollection 2016. PMID 27099761